CLINICAL TRIAL: NCT00856609
Title: The Effects of Exenatide (Byetta) on Energy Expenditure and Weight Loss in Non-Diabetic Obese Subjects
Brief Title: The Effects of Exenatide (Byetta ) on Energy Expenditure and Weight Loss in Nondiabetic Obese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 999909095; 09-DK-N095
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2018-01-19

CONDITIONS: Weight Loss; Obesity
Keywords: Weight Loss; Byetta (Exenatide); Energy Expenditure; Food Intake; Obesity
MeSH Terms: conditions — Weight Loss; Obesity | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Exenatide (Active Comparator): 10 micrograms subcutaneously twice
  Interventions: Drug: Byetta (exenatide); Behavioral: Weight loss
- Placebo (Placebo Comparator): Twice daily
  Interventions: Other: Metabolic Chamber; Drug: Placebo

INTERVENTIONS:
Drug: Byetta (exenatide) — Exenatide is an injectable medication
  Arms: Exenatide
Behavioral: Weight loss — Because response to weight loss
  Arms: Exenatide
Other: Metabolic Chamber — The subject stays in the small room
  Arms: Placebo
Drug: Placebo
  Arms: Placebo

SUMMARY:
Exenatide is an incretin-like drug that has been approved for treatment of type 2 diabetes; it improves glycemia by increasing insulin and decreasing glucagon secretion by pancreatic islet cells and delaying gastric emptying. This randomized, placebo-controlled study is to evaluate whether exenatide over a 5 week period in non-diabetic obese subjects may lead to weight loss. To control for variability in individual response to weight loss treatment, this study will assess the role of exenatide in changing food intake and energy expenditure as possible sources of weight loss. This study will also evaluate the safety profile of exenatide in non-diabetic obese people. Additional assessments will evaluate changes in body fat and hormones involved in the sensations of hunger and fullness.

DETAILED DESCRIPTION:
Obesity can lead to a number of health problems including diabetes, heart disease, stroke, low back pain, fatty liver disease, and osteoarthritis. The medical treatments currently available for obesity are limited. Exenatide is an injectable medication approved for treatment of type 2 diabetes that causes weight loss in some diabetic subjects. The reasons exenatide is thought to cause weight loss include decreased food intake, increased feelings of fullness and nausea. Because levels of a human gut hormone (glucagon like peptide 1) that is similar to exenatide have been shown to be related to resting energy expenditure, it is also possible that exenatide may have effects on a person s metabolism, a.k.a. energy expenditure, but any effect of exenatide on energy expenditure has yet to be evaluated. Even though exenatide is used to treat diabetes, administration of exenatide to non-diabetic lean individuals did not cause frankly low blood sugars.

The primary goal of this study is to investigate the way in which exenatide given twice a day to obese (BMI >= 30 kg/m^2) people without diabetes might lead to weight loss. Because response to weight loss treatment can be highly variable between individuals, we will look at the role of exenatide in changing food intake and energy expenditure as possible explanations for weight loss. We will also assess the safety profile of exenatide in non-diabetic obese people.

This study will involve the use of exenatide or placebo, determined randomly, in obese individuals without diabetes over a 5 week period. The primary measurements will include effects of exenatide on energy expenditure and food intake. We will also look at changes in body fat and the levels of hormones involved in the sensations of hunger and fullness. We will assess if any exenatide-induced changes can predict which individuals lose weight over the 5 weeks. The safety and side effects of exenatide in non-diabetic individuals during this time will also be determined. Findings from this study would help to determine how exenatide works to cause weight loss in people without diabetes, who might benefit most, and would help to improve understanding of why some people respond better to weight loss treatment than others.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Premenopausal women and men < 55 years of age
* BMI >30 kg/m(2)
* Expressed desire for weight loss
* Stable weight (variation < 2.3 kg within past 6 months)
* Ability to provide informed consent
* Ability to follow verbal and written instructions
* Nonsmoker
* Ability to commute to study site on a regular basis for short outpatient visits over 5 weeks
* For females, use of a medically approved form of contraception. For oral contraceptives, subjects will need to be on an established dose for at least 3 months to ensure stable weight and will be asked not to switch contraceptive methods during study participation.

EXCLUSION CRITERIA:

* Age < 18 years
* Use of other medications to treat obesity including medications obtained over the counter or internet, orlistat (Xenical, Alli), sibutramine (Meridia), topiramate (with or without phentermine (Qsymia), phentermine (Adipex P) or lorcaserin (Belviq) within the past 6 months
* History of an eating disorder including anorexia or bulimia
* History of surgery for the treatment of obesity (gastric banding, gastric bypass)
* Diagnosis of type 1 or type 2 diabetes mellitus according to American Diabetes Association guidelines
* Previous exposure to exenatide
* Uncontrolled hypertension as defined by a blood pressure of 150/90 on two or more occasions or use of antihypertensive medications which may affect energy expenditure including alpha blockers, beta blockers, angiotensin receptor blockers or inhibitors of angiotensin converting enzyme
* Current use of tobacco products, marijuana, amphetamines, cocaine or intravenous drug use
* Chronic ethanol use (> 3 drinks /day)
* Endocrine disorders including hypo or hyperthyroidism (including subclinical disease), Cushing s disease, growth hormone deficiency or other pituitary diseases
* History of pancreatitis
* Personal or family history of multiple endocrine neoplasia (MEN)-2 or medullary thyroid cancer
* History of unresolved gallstones
* Hyperamylasemia
* Fasting triglyceride level greater than or equal to 500
* Gastroparesis
* Inflammatory bowel disease or malabsorption disorders
* Malignancy treated with chemotherapy or radiation within the past 5 years
* Current clinical depression, diagnosis of psychosis or recent use of psychotropic medication
* Pregnancy within past 6 months
* Breastfeeding
* Failure to use medically approved contraceptive methods if subject is female
* Liver function abnormalities (transaminases greater than twice normal)
* Renal insufficiency (creatinine clearance < 50 ml/min)
* History of chronic infection including tuberculosis, coccidiomycoses, lyme disease or HIV infection
* Pulmonary disorders, including chronic obstructive pulmonary disease, which would limit ability to follow the protocol (investigator judgment)
* Cardiovascular disease including history of myocardial infarction, unstable angina or heart failure
* Central nervous system disease, including history of cerebrovascular accidents, dementia, and neurodegenerative disorders
* Weight <450 pounds (maximum weight of the DXA machine as per manufacturer s manual)
* Sensitivity to exenatide or any inert components in its formulation
* Sensitivity to acetaminophen
* Conditions not specifically mentioned above may serve as criteria for exclusion at the discretion of the investigators

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2009-03-03; Primary Completion 2016-09-19 (Actual); Study Completion 2016-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Krakoff, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Buse JB, Klonoff DC, Nielsen LL, Guan X, Bowlus CL, Holcombe JH, Maggs DG, Wintle ME. Metabolic effects of two years of exenatide treatment on diabetes, obesity, and hepatic biomarkers in patients with type 2 diabetes: an interim analysis of data from the open-label, uncontrolled extension of three double-blind, placebo-controlled trials. Clin Ther. 2007 Jan;29(1):139-53. doi: 10.1016/j.clinthera.2007.01.015. PMID 17379054
- [Background] Buse JB, Henry RR, Han J, Kim DD, Fineman MS, Baron AD; Exenatide-113 Clinical Study Group. Effects of exenatide (exendin-4) on glycemic control over 30 weeks in sulfonylurea-treated patients with type 2 diabetes. Diabetes Care. 2004 Nov;27(11):2628-35. doi: 10.2337/diacare.27.11.2628. PMID 15504997
- [Background] Amori RE, Lau J, Pittas AG. Efficacy and safety of incretin therapy in type 2 diabetes: systematic review and meta-analysis. JAMA. 2007 Jul 11;298(2):194-206. doi: 10.1001/jama.298.2.194. PMID 17622601
- [Derived] Hollstein T, Basolo A, Ando T, Votruba SB, Krakoff J, Piaggi P. Urinary Norepinephrine Is a Metabolic Determinant of 24-Hour Energy Expenditure and Sleeping Metabolic Rate in Adult Humans. J Clin Endocrinol Metab. 2020 Apr 1;105(4):1145-56. doi: 10.1210/clinem/dgaa047. PMID 32002540
- [Derived] Stinson EJ, Graham AL, Thearle MS, Gluck ME, Krakoff J, Piaggi P. Cognitive dietary restraint, disinhibition, and hunger are associated with 24-h energy expenditure. Int J Obes (Lond). 2019 Jul;43(7):1456-1465. doi: 10.1038/s41366-018-0305-9. Epub 2019 Jan 16. PMID 30651576
- [Derived] Basolo A, Burkholder J, Osgood K, Graham A, Bundrick S, Frankl J, Piaggi P, Thearle MS, Krakoff J. Exenatide has a pronounced effect on energy intake but not energy expenditure in non-diabetic subjects with obesity: A randomized, double-blind, placebo-controlled trial. Metabolism. 2018 Aug;85:116-125. doi: 10.1016/j.metabol.2018.03.017. Epub 2018 Mar 26. PMID 29596853

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 150 planned total number of enrollment, 145 participants were recruited. Among the 145 participants, 84 participants met inclusion criteria. Only 80 participants out of 84 were randomized.
Groups:
- Placebo: Twice daily
  Metabolic Chamber: The subject stays in the small room
  Placebo
Period: Overall Study
Arm/Group | Exenatide | Placebo
Started | 41 | 39
Completed | 40 | 39
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide | Placebo | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (8.4) | 33.7 (9.0) | 34.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 17 | 16 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1 | 9 | 10
  White | 11 | 10 | 21
  Hispanic | 4 | 6 | 10
  Native American | 22 | 14 | 36
  Other | 2 | 0 | 2
Body weight [Mean (Standard Deviation); unit: kg] | 105.5 (19.2) | 108.8 (20.7) | 107.1 (19.9)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 38.0 (6.6) | 38.2 (6.8) | 38.1 (6.7)
Fat free mass [Mean (Standard Deviation); unit: Kg] | 34.6 (11.5) | 37.9 (8.7) | 36.3 (12.8)
Fat mass [Mean (Standard Deviation); unit: Kg] | 27.9 (8.8) | 30.8 (8.7) | 29.4 (8.8)
Body fat [Mean (Standard Deviation); unit: percent] | 44.0 (6.9) | 44.4 (8.7) | 44.2 (7.8)
Fasting glucose [Mean (Standard Deviation); unit: mg/dl] | 96.9 (8.5) | 98.8 (8.8) | 97.8 (8.6)
Two-hour glucose [Mean (Standard Deviation); unit: mg/dl] | 139.4 (25.7) | 135.1 (25.6) | 137.2 (25.6)
Mean energy intake [Mean (Standard Deviation); unit: kcal/day] | 3495.5 (1169.6) | 3093.5 (992.3) | 3294.5 (1096.3)
Percentage of calories needed for weight maintenance participants consumed [Mean (Standard Deviation); unit: Percentage of Carlories] | 119.3 (42.1) | 105.4 (29.6) | 112.3 (36.9)
Carbohydrates intake [Mean (Standard Deviation); unit: kcal/day] | 1785.5 (595.5) | 1593.8 (476.1) | 1689.7 (544.0)
Fat intake [Mean (Standard Deviation); unit: kcal/day] | 1305.3 (488.4) | 1130.9 (484.6) | 1218.1 (491.2)
Protein intake [Mean (Standard Deviation); unit: kcal/day] | 434.2 (159.5) | 396.9 (139.6) | 415.6 (150.1)
Soda intake [Mean (Standard Deviation); unit: kcal/day] | 206.5 (191.3) | 183.3 (169.1) | 195.0 (159.5)
24 hour energy expenditure [Mean (Standard Deviation); unit: kcal/day] | 2319.3 (377.0) | 2333.8 (422.0) | 2325.9 (385.3)
Respiratory quotient [Mean (Standard Deviation); unit: ratio] | 0.86 (0.03) | 0.85 (0.03) | 0.86 (0.03)
Carbohydrate oxidation [Mean (Standard Deviation); unit: kcal/day] | 1121.1 (353.5) | 1068.4 (322.5) | 1097.0 (338.3)
Lipid Oxidation [Mean (Standard Deviation); unit: kcal/day] | 781.0 (330.2) | 873.5 (377.6) | 823.3 (353.1)
Sleeping metabolic rate [Mean (Standard Deviation); unit: kcal/day] | 1818.1 (277.5) | 1800.6 (286.5) | 1810.1 (279.7)
Awake fed thermogenesis [Mean (Standard Deviation); unit: kcal/day] | 629.9 (176.3) | 671.0 (232.0) | 648.7 (203.2)
Spontaneous physical activity [Mean (Standard Deviation); unit: kcal/day] | 80.4 (47.1) | 79.4 (43.4) | 80.0 (45.1)

OUTCOME MEASURES:

1. Primary Outcome: Energy Intake
Description: Mean of 3-day food intake change between 3 days (Day 6-7-8) at baseline assessment and 3 days (Day 12-13-14) during the intervention period between the exenatide and placebo groups
Time Frame: Day 6-7-8 (at baseline) and Day 12-13-14 (3 days after starting study intervention)
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 39 | 39
kcal/day | 1016.1 (724.5) | 245.1 (710.5)
Statistical Analysis 1: Comparison: Exenatide vs Placebo; Test type: Other; p = 0.01, ANCOVA; Slope = -624.8, 95% CI 2-sided [-901.8 to -347.8]

2. Primary Outcome: Twenty-four-hour Energy Expenditure
Description: Change of twenty-four-hour energy expenditure between at Day 5 at baseline assessment and at Day 11 two days after starting study medication between the exenatide and placebo groups
Time Frame: Day 5 and Day 11
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 38 | 33
kcal/day | 51.6 (157.2) | 28.9 (119.7)
Statistical Analysis 1: Comparison: Exenatide vs Placebo; Test type: Other; p = 0.01, ANCOVA; Slope = -24, 95% CI 2-sided [-89.7 to 41.4]

3. Secondary Outcome: Body Weight
Description: Mean decrease between pre- and post-randomization in 5 Weeks between the exenatide and placebo groups.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 31 | 33
kg | 1.6 (3.15) | 0.27 (2.96)
Statistical Analysis 1: Comparison: Exenatide vs Placebo; Test type: Other; p = 0.05, ANCOVA; Slope = -1.48, 95% CI 2-sided [-3.02 to 0.05]

ADVERSE EVENTS:
Arm/Group | Exenatide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 39/40 | 39/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide (N=40) | Placebo (N=39)
hypoglycemia (Endocrine disorders) | 10 | 3
Itchiness (Skin and subcutaneous tissue disorders) | 12 | 4
hunger decrease (Metabolism and nutrition disorders) | 39 | 4
Injection site reaction (Product Issues) | 13 | 5
Nausea (Gastrointestinal disorders) | 24 | 19
Diarrhea (Gastrointestinal disorders) | 16 | 16
Gastroesophageal reflux (Gastrointestinal disorders) | 13 | 15
Headache (General disorders) | 23 | 21
Vomiting (Gastrointestinal disorders) | 11 | 8
Constipation (Gastrointestinal disorders) | 14 | 9
Skin rash (Skin and subcutaneous tissue disorders) | 6 | 1
Palpitations (General disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No